CLINICAL TRIAL: NCT02239510
Title: A Randomized, Double-Blind, Trial Comparing the Efficacy of Linaclotide to Senna in Relieving Symptoms in Patients With Chronic Idiopathic Constipation (CIC)
Brief Title: Efficacy of Linaclotide to Senna for CIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not sufficient recruitment
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14040
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2018-10

CONDITIONS: Chronic Idiopathic Constipation
Keywords: constipation; bowel habits
MeSH Terms: conditions — Constipation | interventions — Sennosides; linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Senna (Active Comparator): 1 capsule (50 mg) Senna daily for 12 weeks
  Interventions: Drug: Senna
- Linzess (Active Comparator): 1 capsule (145 mcg) once daily for 12 weeks
  Interventions: Drug: Linzess

INTERVENTIONS:
Drug: Senna — 1 capsule (50 mg) Senna daily for 12 weeks
  Other Names: sennoside
  Arms: Senna
Drug: Linzess — 1 capsule (145 mcg) of Linzess once daily for 12 weeks
  Other Names: Linaclotide
  Arms: Linzess

SUMMARY:
In this prospective, randomized, double blind study, the aim is to determine the efficacy of Linaclotide in relation to Senna in relieving the symptoms of chronic idiopathic constipation (CIC). Patients with CIC, (age 18 - 70) will be enrolled in the study and randomized to Senna or Linaclotide. Patients will be asked to complete questionnaires during the study and will be followed for 12 weeks. Main outcomes include number of daily bowel movements and measures from surveys regarding bowel habits, relief, and satisfaction.

DETAILED DESCRIPTION:
In this prospective, randomized, double blind study, the aim is to determine the efficacy of Linaclotide in relation to Senna in relieving the symptoms of chronic idiopathic constipation (CIC). Our hypothesis is that Senna is not inferior to Linaclotide in the treatment of CIC. Seventy patients aged 18-70 diagnosed with CIC and seen by a gastroenterologist affiliated with TriHealth or a patient of the Faculty Medical Center clinic will be included in the study. After enrollment, subjects will be randomized to receive either Linaclotide or Senna over a 12-week period after a 1 week wash-out period. During th study period, subjects will complete a log to record the number of daily bowel movements. The subjects will also complete 3 validated surveys on a weekly basis: Subject's Global Assessment SGA of Relief, Subject's Global Assessment SGA of Bowel Habit, and SGA of Satisfaction with their Bowel Habit. A research nurse will meet with subjects at the beginning of the study and then at 3 monthly visits to administer the study medication and distribute the surveys. The main outcomes measures are change in # of bowel movements and SGA survey scores.

ELIGIBILITY:
Inclusion Criteria:

Males and females 18 - 70 years of age. Diagnosed with CIC according to Rome III criteria. Coherent and mentally competent patient to understand and consent for the trial Unremarkable colonoscopy done in past 5 years

Exclusion Criteria:

Significant diarrhea (defined as loose or watery stool and or more than three bowel movements daily associated with urgency more than 25% of the days in preceding 3 months) Untreated hypothyroidism Organic or structural disease as the cause of patient's symptoms (stricture or tumor) Diseases that affect bowel transit time (Gastroparesis, short bowel syndrome) Evidence of cathartic colon History of alcohol, laxative abuse or illicit drug use Pregnant or lactating women Planning pregnancy or become pregnant during study period Concomitant use of any medication that could alter gastrointestinal motility (Calcium channel blockers, Narcotics, anticholinergics, calcium and aluminium containing antacids, phenothiazines, ferrous sulfate)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohd A AlSamman, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Recruitment was low and therefore results are insufficient to share.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from November 2014 to June 2015. A total of 16 patients were screened and 9 patients were enrolled. 3 patients did not show up to appointments and did not complete the study; 6 patients completed the study.
Pre-assignment Details: 1 week wash-out period after enrollment
Groups:
- Senna: Patients who received Senna
- Lizness: Patients who received Lizness
Period: Overall Study
Arm/Group | Senna | Lizness
Started | 5 | 4
Completed | 3 | 3
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Senna | Linzess | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (14.0) | 58 (10.1) | 54 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Bowel Movements Per Week
Description: Change from before to after in number of weekly bowel movements
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: weekly bowel movements
Arm/Group | Senna | Lizness
Number analyzed (Participants) | 3 | 3
weekly bowel movements | 5 (.7) | 2 (2.6)

2. Secondary Outcome: Number of Participants With Relief
Description: Change from before to after treatment in patient assessment of relief - The Subject's Global Assessment (SGA) of Relief was used to measure this outcome. In evaluating subject's response to SGA of relief, subject's who respond with either "completely relieved" or "considerably relieved" for at least 50% of the weeks at the end point or "somewhat relieved" for 100 % of the weeks at the end point will be considered responders to therapy.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Senna | Lizness
Number analyzed (Participants) | 3 | 3
Participants | 2 | 2

3. Secondary Outcome: Change in Assessment of Bowel Habit
Description: Change from before treatment to after treatment in assessment of bowel habit The Subject's Global Assessment (SGA) of Bowel Habit was used to measure this outcome. Patients were asked how bothersome their constipation was in the past week on a scare from 0 (Absent) to 100 (Very Severe).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Senna | Lizness
Number analyzed (Participants) | 3 | 3
scores on a scale | -.20 (.20) | -.08 (.10)

4. Secondary Outcome: Change in Satisfaction With Bowel Habit
Description: Change from before treatment to after treatment on patient satisfaction with bowel habit The Subject's Global Assessment (SGA) of Satisfaction with Bowel Habit was used to measure this outcome. Patients were asked how satisfied they have been with their bowel habits in the previous week on a scale of 0 (Unsatisfied) to 100 (Very Satisfied).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Senna | Lizness
Number analyzed (Participants) | 3 | 3
scores on a scale | .23 (.32) | .03 (.21)

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Linzess: Patients who received Linzess
Arm/Group | Senna | Linzess
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No